CLINICAL TRIAL: NCT00615017
Title: A Placebo-controlled, Double-blind, Dose-escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics and Pharmacodynamics of Single and Multiple Intravenous Infusions of CytoFab (AZD9773) in Patients With Severe Sepsis
Brief Title: AZD9773 Dose Escalation Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: D0620C00004
Record Dates: First submitted 2008-01-31; First posted 2008-02-14 (Estimated); Results first posted 2013-08-22 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-07

CONDITIONS: Severe Sepsis
Keywords: Sepsis; septic shock; Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Sepsis; Shock, Septic; Systemic Inflammatory Response Syndrome | interventions — AZD9773; CytoFab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- AZD9773 cohort 1 (50 units/kg) (Experimental): AZD9773: single infusion of 50 units/kg
  Interventions: Drug: AZD9773 (CytoFab)
- AZD9773 cohort 2 (250 units/kg) (Experimental): AZD9773: single infusion of 250 units/kg
  Interventions: Drug: AZD9773 (CytoFab)
- AZD9773 cohort 3 (250/50 units/kg) (Experimental): AZD9773: loading infusion of 250 units/kg then 9 maintenance doses of 50 units/kg q12hrs
  Interventions: Drug: AZD9773 (CytoFab)
- AZD9773 cohort 4 (500/100 units/kg) (Experimental): AZD9773: loading infusion of 500 units/kg then 9 maintenance doses of 100 units/kg q12hrs
  Interventions: Drug: AZD9773 (CytoFab)
- AZD9773 cohort 5 (750/250 units/kg) (Experimental): AZD9773: loading infusion of 750 units/kg then 9 maintenance doses of 250 units/kg q12hrs
  Interventions: Drug: AZD9773 (CytoFab)
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD9773 (CytoFab) — intravenous infusions
  Arms: AZD9773 cohort 1 (50 units/kg); AZD9773 cohort 2 (250 units/kg); AZD9773 cohort 3 (250/50 units/kg); AZD9773 cohort 4 (500/100 units/kg); AZD9773 cohort 5 (750/250 units/kg)
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled, multi-center, dose-escalation study to assess the safety, tolerability, Pharmacokinetics and Pharmacodynamics of single and multiple ascending intravenous infusions of CytoFab (AZD9773) in adult patients with severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical evidence of infection requiring treatment with parenteral antibiotics
* Patients must meet multiple Systemic Inflammatory Response Syndrome (SIRS) criteria
* Patients must meet criteria for cardiovascular and/or respiratory dysfunction
* Sepsis (infection plus SIRS criteria) must be present prior to organ dysfunction

Exclusion Criteria:

* Moribund and death is considered imminent, or patient not expected to survive 90 days because of underlying medical condition, or classified as Do Not Resuscitate or Do Not Treat
* Patient cannot attain a MAP >60 mmHg when measured via an arterial line and/or a Systolic Blood Pressure (SBP) >80 mmHg in the presence of vasopressors and iv fluids for a period of ≥2 hours
* Receiving immunosuppressants, or high dose steroids within 2 months of provision of informed consent
* Any history of hypersensitivity reaction to sheep products, latex, papain or papaya, or chymopapain or previously administered antivenom manufactured using ovine serum, digoxin immune fab (DigiFab™ , DIGIBIND® ), crotalidae polyvalent immune fab (ovine) (CroFab™ ), or other sheep derived product.
* Treatment with anti Tumor-Necrosis-Factor (anti-TNF) antibodies within 8 weeks before provision of written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Simonson, MD, Study Director — AstraZeneca; Wayne Dankner, MD, Study Director — Parexel
Locations (26):
- United States (26):
  - Research Site, Birmingham, Alabama
  - Research Site, Newark, Delaware
  - Research Site, Bay Pines, Florida
  - Research Site, Miami, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Oak Park, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Hazard, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Kansas City, Missouri
  - Research Site, Camden, New Jersey
  - Research Site, Newark, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Nashville, Tennessee
  - Research Site, Galveston, Texas
  - Research Site, Houston, Texas

REFERENCES:
- [Derived] Yates JW, Das S, Mainwaring G, Kemp J. Population pharmacokinetic/pharmacodynamic modelling of the anti-TNF-alpha polyclonal fragment antibody AZD9773 in patients with severe sepsis. J Pharmacokinet Pharmacodyn. 2012 Dec;39(6):591-9. doi: 10.1007/s10928-012-9270-4. Epub 2012 Sep 23. PMID 23001587

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on January 18, 2008 and the last patient had their last visit on July 30, 2009. Patients were randomised at 17 centres in the United States of America
Pre-assignment Details: 70 adult patients with severe sepsis, clinical evidence of infection requiring parenteral antibiotics, meeting systemic inflammatory response syndrome criteria, and with cardiovascular/respiratory dysfunction were randomised to receive AZD9773 (2 single dose and 3 multiple dose cohorts) in a double-blind, placebo controlled, dose escalation study
Period: Overall Study
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Started | 8 (Patients received treatment) | 9 (Patients received treatment) | 12 (Patients received treatment) | 10 (Patients received treatment) | 8 (Patients received treatment) | 23 (Patients received treatment)
Completed | 8 (Patient completed the study drug) | 8 (Patient completed the study drug) | 7 (Patient completed the study drug) | 9 (Patient completed the study drug) | 7 (Patient completed the study drug) | 20 (Patient completed the study drug)
Not Completed | 0 | 1 | 5 | 1 | 1 | 3
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 2 | 0 | 1 | 1
Not completed — Sepsis resolved | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Transferred out of Intensive Care Unit | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician discontinued drug | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo | Total
Number analyzed (Participants) | 8 | 9 | 12 | 10 | 8 | 23 | 70
Age Continuous [Mean (Standard Deviation); unit: Year] | 53 (11.8) | 49.7 (15) | 55.1 (10.8) | 53 (17.9) | 63.5 (16.1) | 58.9 (17.4) | 56.1 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 7 | 7 | 6 | 12 | 38
  Male | 6 | 5 | 5 | 3 | 2 | 11 | 32
Mechanical ventilation [Number; unit: Participants]
  Yes | 7 | 8 | 9 | 8 | 8 | 20 | 60
  No | 1 | 0 | 2 | 1 | 0 | 3 | 7
  Missing | 0 | 1 | 1 | 1 | 0 | 0 | 3
Organ failure site [Number; unit: Participants]
  Cardiovascular | 2 | 2 | 3 | 3 | 2 | 7 | 19
  Pulmonary dysfunction | 2 | 2 | 3 | 1 | 2 | 3 | 13
  Cardiovascular and pulmonary dysfunction | 4 | 5 | 6 | 6 | 4 | 13 | 38
Shock [Number; unit: Participants]
  Yes | 5 | 6 | 9 | 9 | 7 | 20 | 56
  No | 3 | 3 | 3 | 1 | 1 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Creatinine Values
Description: Change in creatinine values from baseline (pre-infusion) to follow-up (28 days after the start of study drug administration) [calculated as Day 28 mean minus baseline mean]. Safety analysis set (ie all patients who started study drug infusion).
Time Frame: End of study (Day 28)
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Mean (Full Range); unit: μmol/L
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 5 | 4 | 7 | 8 | 6 | 15
μmol/L | -78.6 (-239) [-239 to 8] | -196.8 (-681) [-681 to 0] | -25.1 (-126) [-126 to 44] | -10.9 (-68) [-68 to 167] | 159.0 (-89) [-89 to 1087] | -57.4 (-191) [-191 to 18]

2. Primary Outcome: Change From Baseline in Alanine Aminotransferase Values
Description: Change in alanine aminotransferase values from baseline (pre-infusion) to follow-up (28 days after the start of study drug administration) [calculated as Day 28 mean minus baseline mean]. Safety analysis set (ie all patients who started study drug infusion).
Time Frame: End of study (Day 28)
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Mean (Full Range); unit: μkat/L
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 5 | 3 | 7 | 7 | 6 | 15
μkat/L | -0.998 (-3.24) [-3.24 to 0.16] | 0.017 (-0.25) [-0.25 to 0.43] | -3.133 (-20.62) [-20.62 to -0.03] | -0.520 (-2.05) [-2.05 to 0] | -0.825 (-4.53) [-4.53 to 0.38] | -0.111 (-0.79) [-0.79 to 0.20]

3. Primary Outcome: Change From Baseline in Aspartate Aminotransferase Values
Description: Change in aspartate aminotransferase values from baseline (pre-infusion) to follow-up (28 days after the start of study drug administration) [calculated as Day 28 mean minus baseline mean]. Safety analysis set (ie all patients who started study drug infusion).
Time Frame: End of study (Day 28)
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Mean (Full Range); unit: μkat/L
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 5 | 3 | 7 | 7 | 6 | 15
μkat/L | -2.298 (-5.56) [-5.56 to -0.04] | -0.213 (-0.43) [-0.43 to 0.15] | -3.647 (-21.36) [-21.36 to -0.02] | -0.926 (-3.27) [-3.27 to 0.20] | -0.998 (-3.29) [-3.29 to 0.11] | -0.253 (-1.54) [-1.54 to 0.15]

4. Primary Outcome: Change From Baseline in Bilirubin Values
Description: Change in bilirubin values from baseline (pre-infusion) to follow-up (28 days after the start of study drug administration) [calculated as Day 28 mean minus baseline mean]. Safety analysis set (ie all patients who started study drug infusion).
Time Frame: End of study (Day 28)
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Mean (Full Range); unit: μmol/L
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 5 | 3 | 7 | 7 | 6 | 15
μmol/L | -11.30 (-17.1) [-17.1 to -5.2] | -13.10 (-34.2) [-34.2 to 0] | -10.04 (-49.6) [-49.6 to 0] | -23.71 (-71.8) [-71.8 to 0] | -2.58 (-29.1) [-29.1 to 30.8] | -10.00 (-37.6) [-37.6 to 4.2]

5. Primary Outcome: Change From Baseline in Haemoglobin Values
Description: Change in haemoglobin values from baseline (pre-infusion) to follow-up (28 days after the start of study drug administration) [calculated as Day 28 mean minus baseline mean]. Safety analysis set (ie all patients who started study drug infusion).
Time Frame: End of study (Day 28)
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Mean (Full Range); unit: g/L
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 5 | 4 | 6 | 4 | 5 | 13
g/L | 7 (-18) [-18 to 31] | -16.3 (-42) [-42 to 21] | -0.8 (-31) [-31 to 33] | 6.5 (-5) [-5 to 17] | -13.8 (-35) [-35 to 4] | -4.5 (-47) [-47 to 32]

6. Primary Outcome: Change From Baseline in White Blood Cell Values
Description: Change in white blood cell values from baseline (pre-infusion) to follow-up (28 days after the start of study drug administration) [calculated as Day 28 mean minus baseline mean]. Safety analysis set (ie all patients who started study drug infusion).
Time Frame: End of study (Day 28)
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Mean (Full Range); unit: 10^9 cells/L
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 5 | 4 | 6 | 4 | 5 | 13
10^9 cells/L | -17.552 (-46.67) [-46.67 to -6.11] | -8.975 (-22.58) [-22.58 to 2.18] | 0.413 (-8.11) [-8.11 to 14.84] | -0.225 (-5.60) [-5.60 to 2.86] | -3.482 (-13.42) [-13.42 to 5.82] | -9.987 (-26.40) [-26.40 to 3.34]

7. Primary Outcome: Change From Baseline in Platelet Count Values
Description: Change in platelet count values from baseline (pre-infusion) to follow-up (28 days after the start of study drug administration) [calculated as Day 28 mean minus baseline mean]. Safety analysis set (ie all patients who started study drug infusion).
Time Frame: End of study (Day 28)
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Mean (Full Range); unit: 10^9/L
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 5 | 3 | 5 | 4 | 4 | 13
10^9/L | 287 (-41) [-41 to 650] | 117.3 (18) [18 to 176] | 162 (-56) [-56 to 474] | 72.3 (-114) [-114 to 159] | 252.5 (40) [40 to 591] | 145.1 (-232) [-232 to 735]

8. Primary Outcome: Change From Baseline in Prothrombin Time Values
Description: Change in prothrombin time values from baseline (pre-infusion) to Day 7 [calculated as Day 7 mean minus baseline mean]. Safety analysis set (ie all patients who started study drug infusion).
Time Frame: Day 7
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Mean (Full Range); unit: sec
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 5 | 4 | 6 | 7 | 5 | 17
sec | -3.20 (-8.6) [-8.6 to 2.2] | 0.53 (-0.8) [-0.8 to 2.2] | -1.00 (-2.4) [-2.4 to 0] | -5.31 (-14.7) [-14.7 to 0.4] | 4.36 (-23.8) [-23.8 to 49.4] | 1.68 (-7.5) [-7.5 to 32]

9. Primary Outcome: Change From Baseline in Troponin I
Description: Change in troponin I values from baseline (pre-infusion) to Day 6 [calculated as Day 6 mean minus baseline mean]. Safety analysis set (ie all patients who started study drug infusion).
Time Frame: Day 6
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Mean (Full Range); unit: μg/L
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 8 | 3 | 4 | 9 | 3 | 19
μg/L | -16.454 (-127.37) [-127.37 to 0.26] | -9.523 (-28.58) [-28.58 to 0.01] | -0.630 (-1.61) [-1.61 to 0.10] | -1.434 (-7.21) [-7.21 to 0.04] | -0.027 (-0.07) [-0.07 to 0] | -0.735 (-6.77) [-6.77 to 3.68]

10. Primary Outcome: Change From Baseline in QT With Fridericia Correction (QTcF), Where QT is Measured by ECG, and is the Time Interval Between the Start of the Q Wave and the End of the T Wave in the Heart's Electrical Cycle.
Description: Change in QTcF from baseline (pre-infusion) to Day 1 (end of infusion) for Cohorts 1 and 2 [calculated as Day 1 mean minus baseline mean] and Day 5 (end of infusion) for Cohorts 3 to 5 and placebo [calculated as Day 5 mean minus baseline mean]. Safety analysis set (ie all patients who started study drug infusion).
Time Frame: Day 1 (end of infusion) for Cohorts 1 and 2; Day 5 (end of infusion) for Cohorts 3 to 5 and placebo
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Mean (Full Range); unit: msec
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 7 | 9 | 6 | 9 | 6 | 13
msec | -9.9 (-37) [-37 to 9] | 3.6 (-35) [-35 to 63] | -21.5 (-43) [-43 to -1] | -9.2 (-47) [-47 to 44] | 21.4 (-32) [-32 to 66] | -3.4 (-61) [-61 to 29]

11. Primary Outcome: Change From Baseline in Calculated Mean Arterial Blood Pressure
Description: Change in calculated mean arterial pressure from baseline (pre-infusion) to Day 14 [calculated as Day 14 mean minus baseline mean]. Safety analysis set (ie all patients who started study drug infusion).
Time Frame: Day 14
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Mean (Full Range); unit: mmHg
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 5 | 11
mmHg | 20 (3) [3 to 32] | 7.3 (2) [2 to 13] | 5.3 (-19) [-19 to 34] | 28.7 (4) [4 to 65] | 6.8 (-9) [-9 to 22] | 18 (-4) [-4 to 44]

12. Primary Outcome: Change From Baseline in Body Weight
Description: Change in body weight from baseline (pre-infusion) to Day 6 [calculated as Day 6 mean minus baseline mean]. Safety analysis set (ie all patients who started study drug infusion).
Time Frame: Day 6
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Mean (Full Range); unit: kg
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 7 | 6 | 3 | 5 | 5 | 12
kg | 1.3 (-2) [-2 to 9] | 0.2 (-7) [-7 to 10] | 4 (1) [1 to 8] | 7.4 (-10) [-10 to 25] | 0.2 (-11) [-11 to 14] | 9.9 (0) [0 to 35]

13. Secondary Outcome: 28-Day Mortality
Description: The number of patients who had died at Day 28. Safety analysis set (ie all patients who started study drug infusion).
Time Frame: End of study (Day 28)
Measure: Number; unit: Participants
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 8 | 9 | 12 | 10 | 8 | 23
Participants | 2 | 4 | 5 | 1 | 1 | 6

14. Secondary Outcome: Change From Baseline in Sequential Organ Failure Assessment (SOFA) Scores
Description: Change in SOFA (Sequential Organ Failure Assessment) scores from baseline (pre-infusion) to Day 6 [calculated as Day 6 mean minus baseline mean]. The SOFA score is out of a maximum of 24 (units on a scale 0 to 24). The higher the score, the worse the organ system functioning. Safety analysis set (ie all patients who started study drug infusion).
Time Frame: Day 6
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Mean (Full Range); unit: units on a scale (0 to 24)
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 2 | 3 | 3 | 6 | 3 | 9
units on a scale (0 to 24) | -6 (-7) [-7 to -5] | -2 (-5) [-5 to 0] | -3.3 (-5) [-5 to -2] | -3 (-7) [-7 to 7] | -6 (-11) [-11 to -2] | -4.3 (-8) [-8 to 2]

15. Secondary Outcome: Area Under the Serum Concentration-time Curve From 0 to 12 Hours (AUC(0-12)) of Single Dose AZD9773 Serum Total Fabs (Cohorts 1 and 2)
Description: AUC(0-12) for single dose AZD9773 serum total Fabs (cohorts 1 and 2). PK analysis set (ie a subset of the safety analysis set including only those patients without important deviations that could affect the PK).
Time Frame: Day 1 [PK samples taken pre-dose, the end of each infusion rate and then at 0.5, 1, 2, 8, and 12h post-(last) infusion]
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Geometric Mean (Full Range); unit: μg.h/mL
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 7 | 8 | 0 | 0 | 0 | 0
μg.h/mL | 125.22 [68.6 to 545.3] | 581.01 [197.6 to 1561.8] |  |  |  |

16. Secondary Outcome: Terminal Half-life (t1/2) of Single Dose AZD9773 Serum Total Fabs (Cohorts 1 and 2)
Description: t1/2 of single dose AZD9773 serum total Fabs (cohorts 1 and 2). PK analysis set (ie a subset of the safety analysis set including only those patients without important deviations that could affect the PK).
Time Frame: Day 1 [PK samples taken pre-dose, the end of each infusion rate and then at 0.5, 1, 2, 8, 12, 24, 48, and 72 h post-(last) infusion]
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Mean (Full Range); unit: Hours
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 7 | 6 | 0 | 0 | 0 | 0
Hours | 17.97 (7.8) [7.8 to 30.1] | 19.76 (10.5) [10.5 to 25.6] |  |  |  |

17. Secondary Outcome: Total Apparent Clearance (CL) of Single Dose AZD9773 Serum Total Fabs (Cohorts 1 and 2)
Description: CL of single dose AZD9773 serum total Fabs (cohorts 1 and 2). PK analysis set (ie a subset of the safety analysis set including only those patients without important deviations that could affect the PK).
Time Frame: as for outcome 16
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Mean (Full Range); unit: mL/min/kg
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 7 | 6 | 0 | 0 | 0 | 0
mL/min/kg | 6.11 (1.2) [1.2 to 11.5] | 7.61 (0.8) [0.8 to 16.7] |  |  |  |

18. Secondary Outcome: AUC(0-12) of Loading Dose AZD9773 Serum Total Fabs (Cohorts 3, 4 and 5)
Description: AUC(0-12) of loading dose AZD9773 serum total Fabs (cohorts 3, 4 and 5). PK analysis set (ie a subset of the safety analysis set including only those patients without important deviations that could affect the PK).
Time Frame: Day 1 [PK samples taken pre-dose, the end of each infusion rate and then at 0.5, 1, 2, 8 and 12 h post-(last) infusion]
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Geometric Mean (Full Range); unit: μg.h/mL
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 8 | 9 | 5 | 0
μg.h/mL |  |  | 449.18 [230.2 to 828.8] | 691.53 [474.6 to 1024.7] | 1872.73 [1391.2 to 2559] |

19. Secondary Outcome: Maximum (End of Infusion) Serum Concentration (Cinf) of Loading Dose AZD9773 Serum Total Fabs (Cohorts 3,4 and 5)
Description: Cinf of loading dose AZD9773 serum total Fabs (cohorts 3, 4 and 5). PK analysis set (ie a subset of the safety analysis set including only those patients without important deviations that could affect the PK).
Time Frame: Day 1 [PK samples taken pre-dose, the end of each infusion rate and then at 0.5, 1, 2, 8 and 12 h post-(last)infusion]
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Geometric Mean (Full Range); unit: μg/mL
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 8 | 9 | 5 | 0
μg/mL |  |  | 107.84 [72.3 to 197] | 160.09 [130 to 208] | 351.52 [286 to 443] |

20. Secondary Outcome: Time to Reach Cinf (Tmax) of Loading Dose AZD9773 Serum Total Fabs (Cohorts 3, 4 and 5)
Description: tmax of loading dose AZD9773 serum total Fabs (cohorts 3, 4 and 5). PK analysis set (ie a subset of the safety analysis set including only those patients without important deviations that could affect the PK).
Time Frame: Day 1 [PK samples taken pre-dose, the end of each infusion rate and then at 0.5, 1, 2, 8 and 12 h post-(last)infusion]
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Median (Full Range); unit: Hours
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 8 | 9 | 5 | 0
Hours |  |  | 0.92 [0.5 to 1.4] | 1.08 [0.9 to 1.7] | 1.12 [1.1 to 1.3] |

21. Secondary Outcome: AUC(0-12) of Maintenance Dose AZD9773 Serum Total Fabs (Cohorts 3, 4 and 5)
Description: AUC(0-12) of maintenance dose AZD9773 serum total Fabs (cohorts 3, 4 and 5). PK analysis set (ie a subset of the safety analysis set including only those patients without important deviations that could affect the PK).
Time Frame: PK samples taken pre-dose of Doses 5,7 and 9, then at 0, 0.5, 1, 2, 8 and 12 h post dose 9 infusion
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Geometric Mean (Full Range); unit: μg.h/mL
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 6 | 7 | 4 | 0
μg.h/mL |  |  | 162.82 [66.3 to 440.4] | 251.59 [102.4 to 531.7] | 980.95 [646 to 1524.2] |

22. Secondary Outcome: Cinf of Maintenance Dose AZD9773 Serum Total Fabs (Cohorts 3, 4 and 5)
Description: Cinf of maintenance dose AZD9773 serum total Fabs (cohorts 3, 4 and 5). PK analysis set (ie a subset of the safety analysis set including only those patients without important deviations that could affect the PK).
Time Frame: PK samples taken pre-dose of Doses 5,7 and 9, then at 0, 0.5, 1, 2, 8 and 12 h post dose 9 infusion
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Geometric Mean (Full Range); unit: μg/mL
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 6 | 7 | 4 | 0
μg/mL |  |  | 28.37 [14.6 to 58.4] | 42.51 [8.9 to 71.1] | 151.76 [129 to 184] |

23. Secondary Outcome: Tmax of Maintenance Dose AZD9773 Serum Total Fabs (Cohorts 3, 4 and 5)
Description: tmax of maintenance dose AZD9773 serum total Fabs (cohorts 3, 4 and 5). PK analysis set (ie a subset of the safety analysis set including only those patients without important deviations that could affect the PK).
Time Frame: PK samples taken pre-dose of Doses 5,7 and 9, then at 0, 0.5, 1, 2, 8 and 12 h post dose 9 infusion
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Median (Full Range); unit: Hours
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 0 | 0 | 6 | 7 | 4 | 0
Hours |  |  | 0.54 [0.0 to 0.7] | 1.00 [0.4 to 8.5] | 0.74 [0.5 to 1.6] |

24. Secondary Outcome: Number of Patients Below Tumour Necrosis Factor (TNF)-Alpha Limit of Quantification (LOQ) at 24 Hours (n< LOQ)
Description: Number of patients below tumour necrosis factor (TNF)-alpha limit of quantification (LOQ) at 24 hours (n< LOQ) measured by ELISA (LOQ = 1.3 pg/mL). Safety analysis set (ie all patients who started study drug infusion).
Time Frame: 24 hours
Population: Participants analyzed relates to the number of evaluable patients at the specified time point.
Measure: Number; unit: Participants
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Number analyzed (Participants) | 7 | 9 | 10 | 9 | 5 | 22
Participants | 1.0 | 3.0 | 5.0 | 6.0 | 4.0 | 0.0

ADVERSE EVENTS:
Arm/Group | AZD9773 Cohort 1 (50 Units/kg) | AZD9773 Cohort 2 (250 Units/kg) | AZD9773 Cohort 3 (250/50 Units/kg) | AZD9773 Cohort 4 (500/100 Units/kg) | AZD9773 Cohort 5 (750/250 Units/kg) | Placebo
Serious Adverse Events (participants affected / at risk) | 3/8 | 6/9 | 7/12 | 3/10 | 4/8 | 13/23
Other Adverse Events (participants affected / at risk) | 8/8 | 8/9 | 11/12 | 7/10 | 7/8 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9773 Cohort 1 (50 Units/kg) (N=8) | AZD9773 Cohort 2 (250 Units/kg) (N=9) | AZD9773 Cohort 3 (250/50 Units/kg) (N=12) | AZD9773 Cohort 4 (500/100 Units/kg) (N=10) | AZD9773 Cohort 5 (750/250 Units/kg) (N=8) | Placebo (N=23)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shock Haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Enterocutaneous Fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal Ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical Device Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage Intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxic Epidermal Necrolysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9773 Cohort 1 (50 Units/kg) (N=8) | AZD9773 Cohort 2 (250 Units/kg) (N=9) | AZD9773 Cohort 3 (250/50 Units/kg) (N=12) | AZD9773 Cohort 4 (500/100 Units/kg) (N=10) | AZD9773 Cohort 5 (750/250 Units/kg) (N=8) | Placebo (N=23)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 2 (3) | 4 (4)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leucocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Heparin-Induced Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Atrial Flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 3
Bundle Branch Block Right (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Adrenal Insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Scleral Haemorrhage (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0
Scleral Oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Abdominal Compartment Syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 4
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 3
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 2 | 1 | 0 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Intestinal Ischaemia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 2
General Oedema (General disorders) | 0 | 1 | 3 | 2 | 3 | 3
Asthenia (General disorders) | 1 | 0 | 0 | 1 | 1 | 1
Hypothermia (General disorders) | 0 | 0 | 2 | 0 | 1 | 0
Oedema Periheral (General disorders) | 2 | 0 | 0 | 0 | 1 | 4
Chest Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Face Oedema (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Multi-Organ Failure (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 1 | 1 | 0 | 4
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Ischaemic Hepatitis (Hepatobiliary disorders) | 1 | 0 | 1 | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Enterobacter Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Infected Skin Ulcer (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pelvic Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Systemic Candida (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary Tract Infection Enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Candiduria (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Central Line Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Clostridial Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fungal Skin Infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Herpes Simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lung Infection Pseudomonal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Pneumonia Bacterial (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1
Pneumonia Escherichia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia Staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Bloody Airway Discharge (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Procedural Hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Endotracheal Intubation Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Airway Peak Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood Albumin Decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood Alkaline Phosphatase Decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood Phosphorus Decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood Sodium Decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Brain Natriuretic Peptide Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Breath Sounds Abnormal (Investigations) | 0 | 1 | 1 | 0 | 0 | 2
Clostridium Difficile Toxin Test Positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Ejection Fraction Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Fibrin D Dimer Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Oxygen Saturation Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Troponin Increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Urinary Sediment Present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Urine Output Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 4 | 3 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 3 | 2 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 2 | 1 | 2
Feeding Disorder (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 1
Fluid Overload (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 2 | 0 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lactic Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 2
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Depressed Level Of Consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1
Unresponsive To Stimuli (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 2 | 2 | 1 | 3 | 1 | 4
Anxiety (Psychiatric disorders) | 1 | 0 | 2 | 0 | 1 | 2
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 1 | 0 | 2
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Scrotal Oedema (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 3
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0 | 3
Respiratory Alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0 | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 1 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 6
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1 | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 1 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Periorbital Oedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 2 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 2 | 1 | 1 | 2
Peripheral Coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less